CLINICAL TRIAL: NCT01016184
Title: Prospective, Randomized, Double Blind Placebo Controled Clinical Trial to Assess the Multi- Systemic Effect of Vitamin D Supplementation on Young Men With Vitamin D Deficiency
Brief Title: Influence of Vitamin D Treatment on Multi-systemic Functions in Young Men With Vitamin D Deficiency Due to Work Conditions
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, rambam56, head of metabolic bone disease unit, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: odds3153
Record Dates: First submitted 2009-11-18; First posted 2009-11-19 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2013-01

CONDITIONS: Vitamin D Deficiency
Keywords: Quality of life
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- vitamin D (Active Comparator)
  Interventions: Dietary Supplement: Vitamin D
- placebo (Active Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D — Oral vitamin D 100,000 IU
  Arms: vitamin D
Dietary Supplement: Placebo — Placebo
  Arms: placebo

SUMMARY:
Vitamin D has multiple systemic effects: bone and calcium metabolism, muscle function, insulin responsiveness, body-composition regulation, cell differentiation, and the immune system. Proper status of vitamin D is found to be related to risk reduction in hypertension, cardiac and vascular diseases, autoimmune diseases, and others. Furthermore, vitamin D supplementation resulted in improved endothelial function. Limited sun exposure may lead to vitamin D deficiency, and it may be assumed that modern life styles lead to a lack of sun exposure. Long work-days may be the primary risk factor for vitamin D deficiency. The purpose of this research is to study the effect of vitamin D treatment on multi systemic functions in young healthy men with vitamin D deficiency due to working conditions.

DETAILED DESCRIPTION:
The study has 2 stages: first stage would be survey of 400 employees, who will fill out a questionnaire to identify occupational and demographic risk factors, a nutritional questionnaire, and data from periodic checkups will be collected. Participants will sign a consent form for vitamin D level determinations, and for freezing blood samples. From this survey, the participants that have vitamin D deficiency (25(OH)D levels < 20 ng/ml) will continue to the second stage of the study - administration of vitamin D or placebo. Participants in the interventional study will sign an additional consent form. Length of follow-up: one year. All parameters will be tested at 0, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men between 20-65 years old
* For stage 2: baseline 25(OH)D levels < 20 ng/ml

Exclusion Criteria:

* Liver dysfunction
* Kidney dysfunction
* Patients with unbalanced chronic diseases
* Regular use of medications that lower serum vitamin D levels, or which interfere with intestinal vitamin D absorption

Ages: 25 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 358 (Actual)
Dates: Start 2009-09; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Serum level of 25(OH)D | 12 months

SECONDARY OUTCOMES:
Blood pressure, Endothelial function, Muscle strength. Quality of life, absence from work Laboratory measures:PTH, P1NP, β-CTx, Inflammation markers (hs-CRP), Fasting glucose levels, Insulin, Lipids profile | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam health care campus, Haifa, Israel